CLINICAL TRIAL: NCT01705847
Title: A Phase 1b Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GS-9820 in Subjects With Lymphoid Malignancies
Brief Title: A Phase 1b Study Evaluating GS-9820 in Subjects With Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-315-0102; 2012-000360-19 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoid Malignancies
Keywords: chronic lymphocytic leukemia (CLL); non-Hodgkin lymphoma (NHL); Hodgkin lymphoma (HL); indolent non-Hodgkin lymphoma (iNHL); diffuse large B-cell lymphoma-activated B-cell (DLBCL-ABC); DLBCL-germinal center B-cell (GCB); mantle cell lymphoma (MCL); GS-9820; phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GS-9820 (Experimental): Participants will be sequentially enrolled at progressively higher dose levels to receive GS-9820 administered twice a day. Escalation will proceed to the maximum tolerated dose (MTD), defined as the highest tested dose associated with a rate of dose-limiting toxicities (DLT) of < 33% during the first 4 weeks of therapy.
  Interventions: Drug: GS-9820

INTERVENTIONS:
Drug: GS-9820 — GS-9820 tablets containing 200 mg of GS-9820 administered orally
  Other Names: CAL-120

SUMMARY:
This study is to determine the appropriate dosing regimen of GS-9820 in subjects with lymphoid malignancies. This is a Phase 1b, open-label, dose-escalation and expansion study evaluating the safety, pharmacokinetics, pharmacodynamics, and antitumor activity of GS-9820.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated recurrent B-cell iNHL, DLBCL, MCL, HL or CLL
* Measurable lymphadenopathy
* Requires therapy

Exclusion Criteria:

* Recent history of a major non-lymphoid malignancy
* Evidence of ongoing infection
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 4 weeks
  MTD will be assessed to determine the appropriate dosing regimens for use in future clinical trials of GS-9820 in subjects with lymphoid malignancies.

SECONDARY OUTCOMES:
Overall safety | Up to 5 years
  Overall safety will be assessed by overall safety profile, enumeration and description of any dose-limiting toxicities, serious adverse events, or adverse events leading to discontinuation of study drug.
Pharmacokinetic parameters of GS-9820 as measured by Cmax, Tmax, Ctrough, and AUC | Baseline to Day 29
  * Cmax is defined as the maximum concentration of drug
  * Tmax is defined as the time of Cmax
  * Ctrough is defined as the trough concentration
  * AUC is defined as the area under the plasma concentration versus time curve
Pharmacodynamics to measure changes in the phosphatidylinositol 3-kinase (P13K) delta pathway activation and changes in plasma concentration of disease-associated chemokines and cytokines | Baseline to Day 29
Tumor control | Up to 5 years
  Tumor control as assessed by overall response rate (ORR), time to response (TTR), duration of response (DOR), progression-free survival (PFS), percent change in lymph node area, lymph node response rate, splenomegaly response rate, ALC response rate, hepatomegaly response rate, platelet response rate, hemoglobin response rate, and neutrophil response rate.
Patient well-being assessed using changes in baseline in HRQL (health related quality of life questionnaire) domain and symptom scores based on the Functional Assessment of Cancer Therapy: Lymphoma (FACT-Lym) | Up to 5 years
Drug exposure | Up to 5 years
  Drug administration for GS-9820 as assessed by prescribing records and GS-9820 compliance as assessed by quantification of used and unused drug.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Adewoye, MD, Study Director — Gilead Sciences
Locations (4):
- Netherlands (4):
  - VU Medical Center (VUmc), Amsterdam
  - Academic Medical Center, Amsterdam
  - St. Antonius Hospital, Nieuwegein
  - Erasmus MC - Daniel den Hoed Cancer Center, Rotterdam